CLINICAL TRIAL: NCT05305508
Title: A Randomized, Placebo-controlled, Double-blind, Monocenter, Phase II Trial to Assess the Efficacy of Calcium Dobesilate (CaD) vs. Placebo on SARS-CoV-2 Viral Load Amongst Outpatients With COVID-19.
Brief Title: Assessment of the Efficacy of Calcium Dobesilate vs. Placebo on SARS-CoV-2 Viral Load Amongst Outpatients With COVID-19.
Acronym: COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hervé SPECHBACH (Other)
Collaborators: OM Pharma SA (Industry)
Responsible Party: Sponsor-Investigator, Hervé SPECHBACH, Principal Investigator, Associate Assistant Physician at Primary Care Medicine department HUG, Geneva University Hospitals, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-00000
Record Dates: First submitted 2022-03-25; First posted 2022-03-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: COVID-19 Virus Disease
Keywords: Calcium Dobesilate; Viral load; COVID-19 symptoms
MeSH Terms: conditions — COVID-19 | interventions — Calcium Dobesilate; Mannitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The central pharmacy of the HUG is responsible for preparation of the randomization list and of the blinding of the study treatments. Randomization will be done in variable-sized blocks (size 4) in random sequence.
  Pharmacists will be un-blinded. Care providers and/or outcome assessors, nurses, clinical research associates, investigators and patients will be blinded. Participants will be allocated to either the treatment group (CaD) or placebo group at Day 1 visit through randomization process, and will be dispensed the full treatment regimen on-site, including instructions on intake and explanations of side-effects.
  The investigators will receive from the central pharmacy of the HUG all the study treatments and the participant's allocated treatment randomization number. Thus, the subjects who meet the eligibility criteria will dynamically be randomized at 1:1 ratio and be assigned either to the CaD or to the placebo arms during Day 1 visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): The comparator (placebo, Mannitol 500 mg) will be administered orally twice a day for 7 days.
  Interventions: Drug: Mannitol
- Calcium Dobesilate (Experimental): The CaD (Calcium Dobesilate 500 mg) will be administered orally twice a day for 7 days.
  Interventions: Drug: Calcium Dobesilate

INTERVENTIONS:
Drug: Calcium Dobesilate — The treatment (CaD, Calcium Dobesilate 500 mg) will be administered orally twice a day for 7 days.
  Other Names: DOXIUM 500, OM Pharma
  Arms: Calcium Dobesilate
Drug: Mannitol — The comparator (placebo, Mannitol 500 mg) will be administered orally twice a day for 7 days.
  Other Names: Placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of CaD in reducing SARS-CoV-2 viral load in non-hospitalized adult patients diagnosed with COVID-19, documented with a positive SARS-CoV-2 PCR and with the occurrence of COVID-19 symptoms.

DETAILED DESCRIPTION:
This study is a phase II, randomized, double-blind, placebo-controlled, monocenter trial. The study will assess the efficacy and safety of CaD compared to placebo in reducing SARS-CoV-2 viral load in non-hospitalized adult patients diagnosed with COVID-19, as well as monitoring symptoms severity, progression of the disease to severe form, and persistence of symptoms.

The treatment period is seven consecutive days, followed by a 12-weeks observational period without treatment administration.

Enrolled patients will be randomized, in a ratio of 1:1 into the following treatment groups: - IMP arm: patients will receive 2 x 2 capsules of Calcium Dobesilate (CaD) 500 mg (total of 2000 mg) daily for seven consecutive days

- Placebo arm: patients will receive 2 x 2 capsules of matching placebo (Mannitol 500 mg) daily for seven consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. Documented COVID-19 diagnosis (SARS-CoV-2 positivity as assessed by PCR) ≤3 days of symptom appearance, with a CT<25.
2. Symptoms related to Day 1 ≤ 5 days.
3. Participant presents at least one of the following acute COVID-19 symptoms: nasal congestion or runny nose, sore throat, headache, myalgia, dry/productive cough, fever, chills, abdominal symptoms (nausea, vomiting, diarrhea, abdominal pain), fatigue, chest pain, palpitations, and shortness of breath.
4. Participant is aged ≥ 16 years of age.
5. Participant has provided an appropriate signed Informed consent.

Exclusion Criteria:

1. Known hypersensitivity or allergy to any of the study products to be administered.
2. Participation in any other investigational device or drug study within 30 days preceding study screening visit.
3. Treatment with Calcium Dobesilate or related molecules (e.g., ethamsylate) within 30 days preceding screening visit, or current treatment with any other investigational agent(s).
4. Breastfeeding, unless If the patient agrees to stop breastfeeding
5. Treatment with any investigational, emergency use authorization-approved, or approved drug for COVID-19, such as, but not limited to: monoclonal antibody treatment, direct or indirect antiviral treatment, and others according to local guidelines.
6. Any kind of disorder or medical conditions that, in the opinion of the investigators, may be associated with increased risk to the participant, may affect patients' compliance, or may interfere with study assessments or outcomes.
7. Inability to follow and comply with study procedures.
8. Participant has hospitalization criteria according to local guidelines (Sat < 95%, RR >25) at the time of screening or is admitted to hospital prior to randomization
9. Participant is, in the opinion of the investigators, likely to deteriorate in the next 24-48h and require hospitalization

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | baseline and day 4
  Reduction from baseline of RT-PCR SARS-CoV-2 viral load at day 4, defined by Polymerase Chain Reaction (PCR) threshold cycles. PCR reaction happens in cycles of amplification. Inclusion criteria to enter in the study is a RT-PCR positive for SARS-CoV-2, which correspond to 25 cycles (or lower) of the RT-PCR test. The participant will be tested at day 4 after treatment to evaluate if the viral load has decreased. To do that, another RT-PCR SARS-CoV-2 will be performed. A higher value of RT-PCR cycles compared to the one obtained when the participat was diagnosed COVID-19 positive, is considered a reduction from baseline.

SECONDARY OUTCOMES:
SARS-CoV-2 Viral Load at day 8 | baseline and day 8
  Reduction from baseline of RT-PCR SARS-CoV-2 viral load at day 8.
SARS-CoV-2 Viral Load negativity | day 4, 8 and 21
  Proportion of patients with viral load negativity or very low viral load (defined by PCR threshold cycles >32) at days 4, 8 and 21.
Symptoms | day 4, 8 and 21
  Time to acute symptom resolution after randomisation to treatment.
  Proportion of participants with acute symptom resolution at days 4, 8, 21.
Symptoms resolution | day 4, 8 and 21
  Proportion of participants with acute symptom resolution at days 4, 8, 21.
Persistent COVID-19 symptoms | day 84
  Proportion of patients with persistent symptoms (≥1 of the following symptoms: fatigue, headache, intermittent fever, palpitations/tachycardia, sleep disturbance, anxiety, blurred vision, depression, brain fog (difficulty concentrating), loss of memory, dizziness, tinnitus (and other hearing issues), altered smell, altered taste, shortness of breath, chest pain, cough, myalgia (and spasms), neuralgias, arthralgia (joint pain), paraesthesia, nausea, vomiting, diarrhea, constipation, abdominal pain, menstrual and period problems as well as new onset of allergies) at day 84 (week 12).
Mental and physical score | baseline and 84
  SF12 score at day 21 and day 84 (week 12) compared to day 1 (baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Hervé SPECHBACH, MD, Principal Investigator — HUG
Locations (1):
- Division and Department of Primary Care Medicine, Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Background] Zhou Y, Yang Q, Chi J, Dong B, Lv W, Shen L, Wang Y. Comorbidities and the risk of severe or fatal outcomes associated with coronavirus disease 2019: A systematic review and meta-analysis. Int J Infect Dis. 2020 Oct;99:47-56. doi: 10.1016/j.ijid.2020.07.029. Epub 2020 Jul 25. PMID 32721533
- [Background] Guan WJ, Liang WH, Zhao Y, Liang HR, Chen ZS, Li YM, Liu XQ, Chen RC, Tang CL, Wang T, Ou CQ, Li L, Chen PY, Sang L, Wang W, Li JF, Li CC, Ou LM, Cheng B, Xiong S, Ni ZY, Xiang J, Hu Y, Liu L, Shan H, Lei CL, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Cheng LL, Ye F, Li SY, Zheng JP, Zhang NF, Zhong NS, He JX; China Medical Treatment Expert Group for COVID-19. Comorbidity and its impact on 1590 patients with COVID-19 in China: a nationwide analysis. Eur Respir J. 2020 May 14;55(5):2000547. doi: 10.1183/13993003.00547-2020. Print 2020 May. PMID 32217650
- [Background] Zaim S, Chong JH, Sankaranarayanan V, Harky A. COVID-19 and Multiorgan Response. Curr Probl Cardiol. 2020 Aug;45(8):100618. doi: 10.1016/j.cpcardiol.2020.100618. Epub 2020 Apr 28. PMID 32439197
- [Background] Amraei R, Rahimi N. COVID-19, Renin-Angiotensin System and Endothelial Dysfunction. Cells. 2020 Jul 9;9(7):1652. doi: 10.3390/cells9071652. PMID 32660065
- [Background] Suschek C, Kolb H, Kolb-Bachofen V. Dobesilate enhances endothelial nitric oxide synthase-activity in macro- and microvascular endothelial cells. Br J Pharmacol. 1997 Dec;122(7):1502-8. doi: 10.1038/sj.bjp.0701512. PMID 9421302
- [Background] Zhou Y, Yuan J, Qi C, Shao X, Mou S, Ni Z. Calcium dobesilate may alleviate diabetes-induced endothelial dysfunction and inflammation. Mol Med Rep. 2017 Dec;16(6):8635-8642. doi: 10.3892/mmr.2017.7740. Epub 2017 Oct 9. PMID 29039485
- [Background] Allain H, Ramelet AA, Polard E, Bentue-Ferrer D. Safety of calcium dobesilate in chronic venous disease, diabetic retinopathy and haemorrhoids. Drug Saf. 2004;27(9):649-60. doi: 10.2165/00002018-200427090-00003. PMID 15230646
- [Background] Rabe E, Ballarini S, Lehr L; Doxium EDX09/01 Study Group. A randomized, double-blind, placebo-controlled, clinical study on the efficacy and safety of calcium dobesilate in the treatment of chronic venous insufficiency. Phlebology. 2016 May;31(4):264-74. doi: 10.1177/0268355515586097. Epub 2015 May 18. PMID 25991692
- [Background] Liu J, Li S, Sun D. Calcium Dobesilate and Micro-vascular diseases. Life Sci. 2019 Mar 15;221:348-353. doi: 10.1016/j.lfs.2019.02.023. Epub 2019 Feb 12. PMID 30769115
- [Background] Fernandez IS, Cuevas P, Angulo J, Lopez-Navajas P, Canales-Mayordomo A, Gonzalez-Corrochano R, Lozano RM, Valverde S, Jimenez-Barbero J, Romero A, Gimenez-Gallego G. Gentisic acid, a compound associated with plant defense and a metabolite of aspirin, heads a new class of in vivo fibroblast growth factor inhibitors. J Biol Chem. 2010 Apr 9;285(15):11714-29. doi: 10.1074/jbc.M109.064618. Epub 2010 Feb 9. PMID 20145243
- [Background] Angulo J, Peiro C, Romacho T, Fernandez A, Cuevas B, Gonzalez-Corrochano R, Gimenez-Gallego G, de Tejada IS, Sanchez-Ferrer CF, Cuevas P. Inhibition of vascular endothelial growth factor (VEGF)-induced endothelial proliferation, arterial relaxation, vascular permeability and angiogenesis by dobesilate. Eur J Pharmacol. 2011 Sep 30;667(1-3):153-9. doi: 10.1016/j.ejphar.2011.06.015. Epub 2011 Jun 22. PMID 21703259
- [Background] Angulo J, Cuevas P, Cuevas B, El Youssef M, Fernandez A, Martinez-Salamanca E, Gonzalez-Corrochano R, Gimenez-Gallego G. Diacetyloxyl derivatization of the fibroblast growth factor inhibitor dobesilate enhances its anti-inflammatory, anti-angiogenic and anti-tumoral activities. J Transl Med. 2015 Feb 1;13:48. doi: 10.1186/s12967-015-0413-4. PMID 25638171
- [Background] Njau F, Shushakova N, Schenk H, Wulfmeyer VC, Bollin R, Menne J, Haller H. Calcium dobesilate reduces VEGF signaling by interfering with heparan sulfate binding site and protects from vascular complications in diabetic mice. PLoS One. 2020 Jan 14;15(1):e0218494. doi: 10.1371/journal.pone.0218494. eCollection 2020. PMID 31935212
- [Background] Yin XX, Zheng XR, Peng W, Wu ML, Mao XY. Vascular Endothelial Growth Factor (VEGF) as a Vital Target for Brain Inflammation during the COVID-19 Outbreak. ACS Chem Neurosci. 2020 Jun 17;11(12):1704-1705. doi: 10.1021/acschemneuro.0c00294. Epub 2020 Jun 2. PMID 32485101
- [Background] Clausen TM, Sandoval DR, Spliid CB, Pihl J, Perrett HR, Painter CD, Narayanan A, Majowicz SA, Kwong EM, McVicar RN, Thacker BE, Glass CA, Yang Z, Torres JL, Golden GJ, Bartels PL, Porell RN, Garretson AF, Laubach L, Feldman J, Yin X, Pu Y, Hauser BM, Caradonna TM, Kellman BP, Martino C, Gordts PLSM, Chanda SK, Schmidt AG, Godula K, Leibel SL, Jose J, Corbett KD, Ward AB, Carlin AF, Esko JD. SARS-CoV-2 Infection Depends on Cellular Heparan Sulfate and ACE2. Cell. 2020 Nov 12;183(4):1043-1057.e15. doi: 10.1016/j.cell.2020.09.033. Epub 2020 Sep 14. PMID 32970989
- [Background] Bermejo-Jambrina M, Eder J, Kaptein TM, van Hamme JL, Helgers LC, Vlaming KE, Brouwer PJM, van Nuenen AC, Spaargaren M, de Bree GJ, Nijmeijer BM, Kootstra NA, van Gils MJ, Sanders RW, Geijtenbeek TBH. Infection and transmission of SARS-CoV-2 depend on heparan sulfate proteoglycans. EMBO J. 2021 Oct 18;40(20):e106765. doi: 10.15252/embj.2020106765. Epub 2021 Sep 23. PMID 34510494
- [Background] Moore JB, June CH. Cytokine release syndrome in severe COVID-19. Science. 2020 May 1;368(6490):473-474. doi: 10.1126/science.abb8925. Epub 2020 Apr 17. No abstract available. PMID 32303591
- [Background] Hoffmann M, Kruger N, Schulz S, Cossmann A, Rocha C, Kempf A, Nehlmeier I, Graichen L, Moldenhauer AS, Winkler MS, Lier M, Dopfer-Jablonka A, Jack HM, Behrens GMN, Pohlmann S. The Omicron variant is highly resistant against antibody-mediated neutralization: Implications for control of the COVID-19 pandemic. Cell. 2022 Feb 3;185(3):447-456.e11. doi: 10.1016/j.cell.2021.12.032. Epub 2021 Dec 24. PMID 35026151
- [Background] Takashita E, Kinoshita N, Yamayoshi S, Sakai-Tagawa Y, Fujisaki S, Ito M, Iwatsuki-Horimoto K, Halfmann P, Watanabe S, Maeda K, Imai M, Mitsuya H, Ohmagari N, Takeda M, Hasegawa H, Kawaoka Y. Efficacy of Antiviral Agents against the SARS-CoV-2 Omicron Subvariant BA.2. N Engl J Med. 2022 Apr 14;386(15):1475-1477. doi: 10.1056/NEJMc2201933. Epub 2022 Mar 9. No abstract available. PMID 35263535
- [Derived] Salamun J, Da Silva T, Ustero P, Gosmain Y, Guessous I, Calmy A, Spechbach H. Study protocol for assessment of the efficacy of calcium dobesilate versus placebo on SARS-CoV-2 viral load in outpatients with COVID-19 (CADOVID study): a randomised, placebo-controlled, double-blind, monocentric phase II trial. BMJ Open. 2024 May 8;14(5):e079574. doi: 10.1136/bmjopen-2023-079574. PMID 38719313
- See also: Compendium.ch — https://compendium.ch/product/19768-doxium-caps-500-mg/mpro.
- See also: Boucau J, Marino C, Regan J, Uddin R, Choudhary MC, Flynn JP, et al. Duration of viable virus shedding in SARS-CoV-2 omicron variant infection. MedRxiv Prepr Serv Health Sci. 2 mars 2022; — https://www.medrxiv.org/content/10.1101/2022.03.01.22271582v1